CLINICAL TRIAL: NCT00764309
Title: An Open Label Study to Evaluate the Safety of Dasatinib in the Treatment of Scleroderma Pulmonary Interstitial Fibrosis
Brief Title: Safety Evaluation of Dasatinib in Subjects With Scleroderma Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-267
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-01

CONDITIONS: Scleroderma
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: dasatinib

INTERVENTIONS:
Drug: dasatinib — Tablets, Oral, 100 mg, once daily, 6 months
  Other Names: Sprycel; BMS 354825

SUMMARY:
The purpose of this study was to evaluate the safety of Dasatininb in the treatment of scleroderma pulmonary interstitial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

Target Population

* meet American College of Rheumatology (ACR) criteria for scleroderma
* have clinical evidence of active skin disease with a skin score of ≥15
* have had the onset of their first non-Raynaud phenomenon feature of SSc no more than 3 years prior to screening
* have evidence of fibrosing alveolitis (active pulmonary fibrosis) manifested by a forced vital capacity (FVC) between 45% and 80% of predicted normal and/or diffusing capacity (DLCO) between 30% and 70% of predicted normal values
* have an abnormal high resolution Computed tomography (CT) scan of the chest/lungs demonstrating typical ground glass changes of alveolitis with background fibrosis
* have adequate renal function- no evidence of renal crisis in the 2 months prior to enrollment and serum creatinine < 3 mg/dL
* for both sexes, must use an acceptable form of birth control
* age ≥ 18

Exclusion Criteria:

* Clinically significant pleural or pericardial effusion in the previous 12 months: Grade 3 or 4. Patients with recent Grade I or II effusions or peripheral edema will be permitted to enter the study
* Clinically significant cardiac disease (New York Heart Association Class III or IV) including preexisting arrhythmia, (such as ventricular tachycardia, ventricular fibrillation, or "Torsade de Pointes"), myocardial infarction, uncontrolled angina within 6 months, congestive heart failure, cardiomyopathy, or pericardial disease
* Clinically-significant coagulation or platelet function disorder (eg, known von Willebrand's disease)
* Abnormal QTcF interval prolonged (> 450 msec) after electrolytes have been corrected on baseline electrocardiogram

Laboratory Test Findings

* Hgb < 10 g/dL; platelet count < 100,000/dL; WBC < 3,000/dL; PMN < 1,000/dL; OR lymphocytes < 350/dL
* The presence of any of the following laboratory findings at screening: positive for antibodies to hepatitis C virus; positive for antibodies to hepatitis B surface antigen (HBsAg); serum bilirubin 2 times normal, Alanine Aminotransferase (ALT), or Aspartate Aminotransferase (AST)> 2.5 times upper limit of normal

Prohibited Treatments and/or Therapies

* use of other immunosuppressive therapies must be discontinued at enrollment, eg methotrexate, azathioprine, cyclophosphamide, mycophenolic acid, mycophenolate mofetil, cyclosporine
* treatment with any other experimental or investigational drug(s) concurrently or less than 12 weeks prior to study enrollment
* use of anti-fibrotic agents must be discontinued at enrollment, eg colchicine, D-penicillamine, minocycline or Type 1 oral collagen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Ucla Division Of Rheumatology, Los Angeles, California
  - University Of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University Feinberg School Of Medicine, Chicago, Illinois
  - Boston University School Of Medicine, Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - West Michigan Rheumatology, Grand Rapids, Michigan
  - Umdnj Clinical Research Center, New Brunswick, New Jersey
  - Hospital For Special Surgery, New York, New York
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University Of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Martyanov V, Kim GJ, Hayes W, Du S, Ganguly BJ, Sy O, Lee SK, Bogatkevich GS, Schieven GL, Schiopu E, Marangoni RG, Goldin J, Whitfield ML, Varga J. Novel lung imaging biomarkers and skin gene expression subsetting in dasatinib treatment of systemic sclerosis-associated interstitial lung disease. PLoS One. 2017 Nov 9;12(11):e0187580. doi: 10.1371/journal.pone.0187580. eCollection 2017. PMID 29121645
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 47 participants enrolled, 31 were treated. Reasons for not entering treatment period were: withdrew consent-1, lost to follow up-2, no longer met study criteria-12, other reasons-1.
Groups:
- 100 mg Dasatinib, Oral Administration: Participants received 100 mg dasatinib once daily orally for up to 2 years (6 months of dosing to evaluate the primary endpoint + 18 months of dosing to assess longer-term safety and efficacy)
Period: Overall Study
Arm/Group | 100 mg Dasatinib, Oral Administration
Started | 31 (Number of participants treated.)
Completed | 31 (Completed=off study. Major Reasons for off study: AE-13; withdrawn by sponsor-10; Lack of efficacy-3)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 100 mg Dasatinib, Oral Administration
Number analyzed (Participants) | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 50.8 (12.44)
Age, Customized [Number; unit: Years]
  <65 years | 26
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 10
Race/Ethnicity, Customized [Number; unit: participants]
  White | 24
  Black / African American | 3
  American Indian/Alaska Native | 1
  Other | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 3
  Not Hispanic/Latino | 28
Baseline Pulmonary Function: Diffusion capacity [Mean (Standard Deviation); unit: mL/min/mmHg] — Diffusing capacity (DLCO) is the carbon monoxide uptake from a single inspiration in a standard time (usually 10 sec).
  There were 29 participants with observations for this measure.
  mL/min/mmHg | 14.223 (4.8012)
Baseline Pulmonary Function [Mean (Standard Deviation); unit: Liters] — Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration; Forced expiratory volume in 1 second (FEV1) is volume that has been exhaled at the first second of forced expiration; Total lung capacity (TLC) is the maximum volume of air present in the lungs.
  n=participants with observations
  Liters
    FVC, n=30 | 2.955 (0.7978)
    FEV1, n=30 | 2.614 (1.3495)
    TLC, n=26 | 4.292 (1.1784)
Time from Initial Scleroderma Diagnosis to Start of Study [Number; unit: Participants]
  < 12 months | 12
  12 - 23 months | 8
  24 - 36 months | 7
  > 36 months | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died, Experienced Serious Adverse Events (SAEs), or Adverse Events (AEs)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug. SAE: any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was an overdose. Participants who discontinued the study due to any AEs were recorded.
Time Frame: From start of study drug therapy up to 30 days after the last dose. The duration of dasatinib dosing in this study was up to 2 years
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | 100 mg Dasatinib, Oral Administration
Number analyzed (Participants) | 31
Participants
  Deaths | 0
  AEs | 31
  SAEs | 7
  Drug-Related Death | 0
  Drug-Related AEs | 24
  Drug-Related SAEs | 5

2. Primary Outcome: Reasons for Discontinuation of Study Treatment
Description: Participants who discontinued the study due to any AEs were recorded.
  Significant drug-related discontinuations were those SAEs recorded on the SAE case report forms with relationship to study drug of related or missing and action taken regarding study drug of discontinued or missing.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | 100 mg Dasatinib, Oral Administration
Number analyzed (Participants) | 31
Participants
  AEs | 13
  SAEs | 4
  Drug-Related AEs | 8
  Drug-Related SAEs | 3
  Significant Drug-Related Pericardial Effusion | 0
  Significant Drug-Related Pleural Effusion | 2
  Significant Drug-Related Bone Marrow Suppression | 0
  Significant Worsening of Underlying Scleroderma | 0
  Unforeseen toxicity of dasatinib | 0
  Significant Drug-Related Peripheral Edema | 0

3. Primary Outcome: Laboratory Test Results Summary of Toxicity: Hematology
Description: Toxicity was graded as per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 3.0. (Grade (GR)0=normal, GR1=mild, GR2=moderate, GR3=severe, GR4=life threatening). Granulocyte count (x 10^9 /L), GR1: ≥1.0 - <1.5, GR2: ≥0.5 - <1.0; Hemoglobin (g/dL), GR0: 13-17, GR1: <13 - 10.0 , GR2: 8.0 - <10.0, GR3: 6.5 - <8.0; Platelet count (x 10^9 /L) GR0: 150-400, GR2: ≥50.0 - <75.0; Leukocyte count (x 10^9 /L ), GR0: 3.5-11.1, GR2: 2.0 - <3.0.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | 100 mg Dasatinib, Oral Administration
Number analyzed (Participants) | 31
participants
  Granulocyte count, GR0 | 28
  Granulocyte count, GR1 | 1
  Granulocyte count, GR2 | 1
  Granulocyte count, GR not reported | 1
  Hemoglobin, GR0 | 4
  Hemoglobin, GR1 | 17
  Hemoglobin, GR2 | 8
  Hemoglobin, GR3 | 1
  Hemoglobin, GR not reported | 1
  Platelet count, GR0 | 29
  Platelet count, GR2 | 1
  Platelet count, GR not reported | 1
  Leukocyte count, GR0 | 29
  Leukocyte count, GR2 | 1
  Leukocyte count, GR not reported | 1

4. Primary Outcome: Laboratory Test Results Summary of Toxicity: Blood Chemistry Per (NCI-CTCAE) Version 3.0 Grade (GR)
Description: GR0=normal,1=mild,2=moderate,3=severe,4=life-threatening. ALP(U/L) GR0:40-135,GR1:>135-337; ALT(U/L) GR0:0-47,GR1:>47-117; AST(U/L) GR0:0-37,GR1:>37-93; High(↑) Calcium(mg/dL) GR0:8.4-10.2,GR1:>10.2-11.5; Low(↓) Calcium(mg/dL) GR0:8.4-10.2,GR1:<8.4-8.0,GR2:7.0-<8.0; CK(U/L) GR0:24-195,GR1:>195-488, GR2:>488-975; Creatinine(mg/dL) GR0:0.6-1.4,GR1:>1.4-2.1,GR2:>2.1-4.2; ↑Potassium(mEq/L) GR0:3.6-5.2,GR1:>5.2-5.5,GR2:>5.5-6.0; ↑Sodium(mEq/L) GR0:134-146; ↓Sodium(mEq/L) GR0:134-146,GR1:<134-130; Inorganic Phosphorus(mg/dL) GR0:2.4-4.9,GR2:≥2.0-<2.5; Total Bilirubin(mg/dL) GR0:0-1.1,GR1:>1.1-2.75.
Time Frame: as for outcome 1
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | 100 mg Dasatinib, Oral Administration
Number analyzed (Participants) | 31
participants
  Alkaline Phosphatase (ALP), GR0 | 30
  ALP, GR1 | 1
  Alanine Aminotransferase (ALT), GR0 | 24
  ALT, GR1 | 7
  Aspartate Aminotransferase (AST), GR0 | 21
  AST, GR1 | 10
  High Calcium, GR0 | 23
  High Calcium, GR1 | 8
  Low Calcium, GR0 | 28
  Low Calcium, GR1 | 2
  Low Calcium, GR2 | 1
  Creatine Kinase (CK), GR0 | 16
  CK, GR1 | 11
  CK, GR2 | 2
  CK, GR not reported | 2
  Creatinine, GR 0 | 26
  Creatinine, GR1 | 3
  Creatinine, GR2 | 2
  High Potassium, GR0 | 28
  High Potassium, GR1 | 2
  High Potassium, GR2 | 1
  Low Potassium, GR 0 | 27
  Low Potassium, GR 1 | 4
  High Sodium, GR0 | 31
  Low Sodium, GR0 | 28
  Low Sodium, GR1 | 3
  Inorganic Phosphorus, GR 0 | 30
  Inorganic Phosphorus, GR 2 | 1
  Total Bilirubin, GR0 | 30
  Total Bilirubin, GR1 | 1

ADVERSE EVENTS:
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 7/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=31)
ATRIAL FLUTTER (Cardiac disorders) | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 1
DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1
FACE OEDEMA (General disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1
CYSTITIS (Infections and infestations) | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1
CLOSTRIDIAL INFECTION (Infections and infestations) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=31)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
DYSPEPSIA (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 8
PRURITUS (Skin and subcutaneous tissue disorders) | 3
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 8
INFLUENZA LIKE ILLNESS (General disorders) | 2
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 3
PARAESTHESIA ORAL (Gastrointestinal disorders) | 2
WEIGHT DECREASED (Investigations) | 3
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2
FLUSHING (Vascular disorders) | 2
HAEMOGLOBIN DECREASED (Investigations) | 3
INSOMNIA (Psychiatric disorders) | 5
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 3
URINARY TRACT INFECTION (Infections and infestations) | 4
CARBON MONOXIDE DIFFUSING CAPACITY DECREASED (Investigations) | 2
DIARRHOEA (Gastrointestinal disorders) | 12
DIZZINESS (Nervous system disorders) | 4
GLOSSODYNIA (Gastrointestinal disorders) | 2
HAEMATOCHEZIA (Gastrointestinal disorders) | 2
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2
SKIN TIGHTNESS (Skin and subcutaneous tissue disorders) | 2
ALOPECIA (Skin and subcutaneous tissue disorders) | 3
BRONCHITIS (Infections and infestations) | 2
CHEST PAIN (General disorders) | 2
INFECTED SKIN ULCER (Infections and infestations) | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2
FATIGUE (General disorders) | 12
FOLLICULITIS (Infections and infestations) | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 2
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4
PYREXIA (General disorders) | 2
RASH (Skin and subcutaneous tissue disorders) | 6
COUGH (Respiratory, thoracic and mediastinal disorders) | 8
HEADACHE (Nervous system disorders) | 8
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2
SINUSITIS (Infections and infestations) | 4
VITAL CAPACITY DECREASED (Investigations) | 2
ANAEMIA (Blood and lymphatic system disorders) | 6
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3
DEPRESSION (Psychiatric disorders) | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 3
OEDEMA PERIPHERAL (General disorders) | 6
PALPITATIONS (Cardiac disorders) | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3
RAYNAUD'S PHENOMENON (Vascular disorders) | 3
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4
VOMITING (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication